CLINICAL TRIAL: NCT05691452
Title: Technology-Based Sedentary Reduction Intervention in Patients With Type 2 Diabetes: A Pilot Study
Brief Title: Technology Based Sedentary Reduction Intervention in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Chorong Park, Assistant Professor, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 221566
Record Dates: First submitted 2023-01-05; First posted 2023-01-20 (Actual); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes; Sedentary Behavior; Physical Activity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): The intervention group will target a 120 minute per day reduction in sedentary behavior using an objective activity monitor and mHealth.
  Interventions: Behavioral: Sit Less Program

INTERVENTIONS:
Behavioral: Sit Less Program — The intervention group will target a 120 minute per day reduction in sedentary behavior using an objective activity monitor and mHealth. Outcomes will be measured at baseline and post-intervention.

SUMMARY:
The purpose of this study is to develop and test an 8-week sedentary behavior reduction intervention ("Sit Less" program) for patients with type 2 diabetes. The program aims to reduce and break sitting times among this population using an objective activity monitor and mHealth. The investigators will test the program to help diabetes patients break up sitting time, reduce daily sitting time, and move more. The investigators will also study preliminary effects of the SB reduction intervention on light physical activity, cardiometabolic markers and patient-centered outcomes, and whether diabetes patients like the program and can follow it.

DETAILED DESCRIPTION:
The investigators propose to develop and conduct a pilot study to test a wearable technology-based sedentary behavior reduction intervention in type 2 diabetes patients. The participants in the first cohort (n=15), 'Sit Less Version 1' will be randomized to either the control group or the sedentary behavior reduction intervention group. The intervention group will target a 120 minute per day reduction in sedentary behavior using an objective activity monitor and mHealth. The study will have an iterative design process with multiple cohorts. After the first cohort completed the study, we will collect their feedback to modify the Sit Less program. With Sit Less Version 2, Cohort 2 (n=20) participants will participate in the intervention as a single group, without randomization. The Sit Less Version 2 will be 8 weeks long.

Specifically, the study aims to: determine the feasibility and acceptability of the sedentary behavior reduction intervention in type 2 diabetes patients by evaluating reach, retention, satisfaction, and compliance with the intervention; evaluate the preliminary efficacy of the sedentary behavior reduction intervention on changes in sedentary time; and explore preliminary effects of the sedentary reduction intervention on physical activity, cardiometabolic markers and patient-centered outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ages 18 and above
* diagnosed with type 2 diabetes
* self-reported HbA1C<13
* self-report of sitting ≥ 8hr/day
* ability to stand and walk
* ownership of a smartphone.

Exclusion Criteria:

* currently using an activity tracker
* use of insulin
* random blood glucose >300
* currently participating in exercise or other research programs
* non-English speaking
* patients who are classified as unstable (e.g. heart failure, uncontrolled arrhythmia) or have kidney disease that limits daily water intake, or any other conditions contradictory to standing or walking
* currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chorong Park, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 - Control: Control Group (n=8) Participants in this group received standard care and did not participate in the "Sit Less" intervention.
- Cohort 1 - Intervention: Sit Less Intervention Group (n=5) Participants in this group received the 8-week "Sit Less" sedentary behavior reduction intervention, which targeted a 120 minute per day reduction in sedentary time using an activity monitor and mHealth tools.
- Cohort 2 - Intervention: Sit Less Intervention Group (n=15) All participants in Cohort 2 received the modified "Sit Less Version 2" sedentary behavior reduction intervention, which was an 8-week program using an activity monitor and mHealth tools to target a reduction in daily sedentary time.
Period: Overall Study
Arm/Group | Cohort 1 - Control | Cohort 1 - Intervention | Cohort 2 - Intervention
Started | 10 | 6 | 15
Completed | 8 | 5 | 13
Not Completed | 2 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline characteristics were reported for each of these three analysis populations (Cohort 1 Control, Cohort 1 Intervention, and Cohort 2 Intervention).
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Control | Cohort 1 - Intervention | Cohort 2 - Intervention | Total
Number analyzed (Participants) | 8 | 5 | 15 | 28
Age, Categorical [Count of Participants; unit: Participants] — Population: The study included a total of 31 participants across 2 cohorts:
  Cohort 1 (n=13) Sit Less Intervention Group (n=5) Control Group (n=8) Cohort 2 (n=15) Sit Less Intervention Group (n=15)
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 5 | 3 | 12 | 20
    >=65 years | 3 | 2 | 3 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.54 (16.67) | 60.54 (16.67) | 57.4 (15.1) | 59.8 (16.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 8 | 17
  Male | 3 | 1 | 7 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 6 | 4 | 12 | 22
  Non-Hispanic Black | 1 | 1 | 2 | 4
  Asian | 1 | 0 | 1 | 2
BMI [Mean (Standard Deviation); unit: kg/m2] | 31.58 (3.98) | 37.46 (5.92) | 32.25 (5.65) | 33.11 (5.40)

OUTCOME MEASURES:

1. Primary Outcome: Level of Satisfaction With the Intervention Assessed by Lyons et al and Burner et al.'s Questionnaires
Description: Acceptability of the Sit Less program will be assessed using satisfaction surveys and exit interviews with Sit Less group participants. The surveys combined items from two questionnaires: Lyons et al., which measured overall program satisfaction (e.g., "I would recommend the program"), ease of use, and intention to continue using each program component, and Burner et al., which evaluated the text messaging component, including content relevance, motivational impact, frequency, and timing. Satisfaction with the overall program will be evaluated with six items like "I would recommend the program" and "The program is likely to reduce sedentary behavior." All responses will be made on a Likert-type scale from 1 (strongly disagree) to 5 (strongly agree). Higher scores mean higher levels of satisfaction.
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cohort 1 - Intervention | Cohort 2 - Intervention
Number analyzed (Participants) | 5 | 13
score on a scale
  I would recommend the program to family and friends. | 5 [3 to 5] | 4 [4 to 5]
  I enjoyed the sedentary behavior reduction program | 5 [2 to 5] | 4 [4 to 5]
  This program is likely to increase awareness of my sedentary behavior | 5 [3.5 to 5] | 5 [4.5 to 5]
  This program is likely to change attitudes toward my sedentary behavior | 5 [3.5 to 5] | 5 [4 to 5]
  This program is likely to increase intentions/motivation to reduce sedentary behavior | 4 [3.5 to 5] | 5 [4 to 5]
  Participation in this program is likely to reduce sedentary behavior | 4 [3.5 to 5] | 5 [4 to 5]
  Fitbit satisfaction | 5 [4 to 5] | 5 [3.5 to 5]
  Satisfaction on smart water bottle satisfaction | 4 [2.5 to 5] | 4 [3 to 4.5]
  Satisfaction on text message satisfaction | 4 [3 to 5] | 3 [2.5 to 4]
  Goal setting was useful | 5 [3 to 5] | 4 [4 to 4]
  Text message timing | 4 [3.5 to 5] | 4 [3 to 4]
  Text message frequency | 4 [3.5 to 5] | 4 [3.5 to 4]

2. Primary Outcome: Level of Compliance With the Intervention Assessed by Number of Days the Fitbit Device Was Worn
Description: The compliance with the intervention will be assessed by number of days the Fitbit device was worn per week.
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: days per week
Arm/Group | Cohort 1 - Intervention | Cohort 2 - Intervention
Number analyzed (Participants) | 5 | 15
days per week | 6.58 [6.13 to 6.94] | 6.13 [5.63 to 7]

3. Primary Outcome: Changes of Total Daily Sedentary Time
Description: Total daily sedentary time will be measured from 7 days of activPAL 3 device monitoring.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Cohort 1 - Control | Cohort 1 - Intervention | Cohort 2 - Intervention
Number analyzed (Participants) | 8 | 5 | 13
minutes
  Baseline | 622.5488 (86.68241) | 670.8750 (99.19531) | 640.7781 (149.77000)
  Post-intervention | 554.6351 (68.21266) | 602.8750 (122.18354) | 609.5371 (155.22499)
Statistical Analysis 1: Comparison: Cohort 1 - Control vs Cohort 1 - Intervention; Test type: Superiority; p = 0.578, Regression, Linear — Generalized linear models generated estimated mean differences in the post-intervention values controlling for the baseline assessments; Mean Difference (Net) = 20.05, 95% CI 2-sided [-50.68 to 90.78]

4. Primary Outcome: Changes of Prolonged Sedentary Time
Description: Prolonged sitting time (time spent sitting >60mins) will be measured by 7 days of activPAL 3 device monitoring.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Cohort 1 - Control | Cohort 1 - Intervention | Cohort 2 - Intervention
Number analyzed (Participants) | 8 | 5 | 13
minutes
  Baseline | 262.978375 (167.0212359) | 226.240200 (97.8064178) | 187.086785 (110.8965832)
  Post-intervention | 198.121663 (140.8557184) | 147.582360 (140.4909207) | 165.056000 (126.7480441)
Statistical Analysis 1: Comparison: Cohort 1 - Control vs Cohort 1 - Intervention; Test type: Superiority; p = 0.61, Regression, Linear; Mean Difference (Net) = -21.2, 95% CI 2-sided [-101.9 to 59.5]

5. Primary Outcome: Changes of Sit-to-stand Transitions
Description: Number of sit-to-stand transitions will be measured by 7 days of activPAL 3 device monitoring.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: Sit-to-Stand Transitions
Arm/Group | Cohort 1 - Control | Cohort 1 - Intervention | Cohort 2 - Intervention
Number analyzed (Participants) | 8 | 5 | 13
Sit-to-Stand Transitions
  Baseline | 31.25 (12.510) | 42.80 (9.445) | 46.08 (19.448)
  Post-intervention | 32.75 (11.298) | 43.20 (8.167) | 45.31 (15.250)
Statistical Analysis 1: Comparison: Cohort 1 - Control vs Cohort 1 - Intervention; Test type: Superiority; p = 0.674, Regression, Linear; Mean Difference (Net) = 1.55, 95% CI 2-sided [-5.68 to 8.78]

6. Secondary Outcome: Changes of Physical Activity Measured by 7 Days of activPAL Device Monitoring
Description: Physical activity will be considered stepping time (minutes), measured by 7 days of activPAL monitoring.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Cohort 1 - Control | Cohort 1 - Intervention | Cohort 2 - Intervention
Number analyzed (Participants) | 8 | 5 | 13
minutes
  Baseline | 37.547425 (19.0937877) | 63.195200 (18.4359097) | 67.806546 (18.0175217)
  Post-intervention | 54.1757038 (29.75937131) | 75.4577200 (60.05685663) | 75.1487769 (24.21793627)
Statistical Analysis 1: Comparison: Cohort 1 - Control vs Cohort 1 - Intervention; Test type: Superiority; p = .013, Regression, Linear; Mean Difference (Net) = -21.6, 95% CI 2-sided [-38.5 to -4.59]

7. Secondary Outcome: Changes of Confidence in Reducing Sedentary Behavior Measured by Using 6 Items From the Self-Efficacy Questionnaire for Physical Activity and Sedentary Behavior.
Description: Confidence in reducing sedentary behavior will be measured using 6 items from the Self-Efficacy Questionnaire for Physical Activity and Sedentary Behavior. The items assess the level of confidence for specific sitting behaviors and sedentary breaks. Each item is a likert-type scale, ranging from 1 to 5. Higher scores mean a better outcome.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 - Control | Cohort 1 - Intervention | Cohort 2 - Intervention
Number analyzed (Participants) | 8 | 5 | 13
score on a scale
  Baseline | 3.9038 (.68874) | 3.7000 (.83666) | 3.9038 (.6887)
  Post-intervention | 3.3750 (1.22474) | 3.8500 (0.89443) | 3.3846 (.89916)
Statistical Analysis 1: Comparison: Cohort 1 - Control vs Cohort 1 - Intervention; Test type: Superiority; p = 0.29, Regression, Linear; Mean Difference (Net) = 0.387, 95% CI 2-sided [-0.335 to 1.109]

8. Secondary Outcome: Changes of Habit Strength for Sedentary Behavior Assessed by Using the Self-Report Habit Index.
Description: Habit strength for sedentary behavior will be assessed by 7 items from the Self-Report Sedentary Behavior Habit Index. This measure will evaluate changes in habit strength for sedentary behavior, assessed using the Self-Report Habit Index adapted for sedentary breaks (standing/walking). Habit strength for sedentary behavior will be assessed by using a validated measure, Self-Report Habit Index (Cronbach's alpha = 0.91). This 7- item index was adapted to sedentary breaks (standing/walking) to assess the degree to which sedentary breaks become habitual. Each item is rated on a 5-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). The total score is calculated by taking the mean of the 7 items, which range from 1 to 7, with higher scores indicating a stronger habit strength for taking sedentary breaks.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 - Control | Cohort 1 - Intervention | Cohort 2 - Intervention
Number analyzed (Participants) | 8 | 5 | 13
score on a scale
  Baseline | 6.2143 (.63430) | 6.0857 (1.18924) | 5.2967 (1.57517)
  Post-intervention | 5.8214 (1.10327) | 5.5143 (1.24786) | 5.8462 (1.02430)
Statistical Analysis 1: Comparison: Cohort 1 - Control vs Cohort 1 - Intervention; Test type: Superiority; p = 0.701, Regression, Linear; Mean Difference (Net) = -0.203, 95% CI 2-sided [-1.24 to 0.833]

9. Secondary Outcome: Changes of 24-hour Mean Glucose Levels Assessed by Continuous Glucose Monitors
Description: 24-hour glucose levels will be measured by the use of a continuous glucose monitor over a 7-day period. The 24-hour glucose control will be evaluated by mean 24-hour glucose levels.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Cohort 1 - Control | Cohort 1 - Intervention | Cohort 2 - Intervention
Number analyzed (Participants) | 7 | 4 | 13
mg/dL
  Baseline | 120.7143 (21.83052) | 135.2500 (29.15905) | 129.3846 (28.43278)
  Post-intervention | 126.0000 (56.60094) | 115.7500 (20.51625) | 153.5385 (35.08945)
Statistical Analysis 1: Comparison: Cohort 1 - Control vs Cohort 1 - Intervention; Test type: Superiority; p = 0.376, Regression, Linear; Mean Difference (Net) = -21.45, 95% CI 2-sided [-68.99 to 26.08]

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: The adverse event data were collected throughout the 8-week study period. The definition of adverse event used in this study is consistent with the clinicaltrials.gov definition - any untoward medical occurrence associated with the use of an intervention, whether or not considered related to the intervention. Serious adverse events, as defined by the FDA, were not observed in this study.
Arm/Group | Cohort 1 - Control | Cohort 1 - Intervention | Cohort 2 - Intervention
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 0/15
Other Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - Control (N=10) | Cohort 1 - Intervention (N=6) | Cohort 2 - Intervention (N=15)
Back pain and anxiety (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Participant DM0027 reported increased back pain and anxiety due to the Sit Less program, leading to their withdrawal on 11/6/2023. The PI was informed and agreed with the withdrawal.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT05691452/Prot_SAP_001.pdf
  • Informed Consent Form (2023-11-10): https://cdn.clinicaltrials.gov/large-docs/52/NCT05691452/ICF_000.pdf